CLINICAL TRIAL: NCT05962853
Title: Effect of Trans Electrical Nerve Stimulation on Patient Outcomes After Laparoscopic Cholecystectomy: A Randomized Controlled Study
Brief Title: Effect of TENS on Patient Outcomes After Laparoscopic Cholecystectomy
Acronym: TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cansel Bozer, specialist nurse, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-02
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cholecystitis; Gallstone; Cholecystolithiasis
Keywords: Pain; Cholecystectomy; Nurse; TENS
MeSH Terms: conditions — Cholecystitis; Gallstones; Cholecystolithiasis; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Application of the experimental group: 2 hours after the surgery, TENS will be applied for 30 minutes and then TENS will be applied 3 times at 8 hour intervals. Postoperatively at the 2nd hour (just before TENS), at the 3rd hour (1 hour after the onset of TENS), at the 10th hour (just before the TENS), at the 11th hour (1 hour after the start of TENS), at the 18th hour ( Just before TENS) at the 19th Hour (1 hour after the start of TENS). In order to protect sleep integrity, TENS application hours will be arranged according to the patient.
  Application of the control group: TENS will not be applied to this group
Who Masked: Participant, Outcomes Assessor
Masking Description: Application will be made by the researcher and the outcome will be assessements will be performed by a investigator who is blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group ( TENS will be applied ) (Experimental): After 30 minutes of TENS application 2 hours after the surgery, TENS will be applied 3 times at 8 hour intervals. Postoperatively at the 2nd hour (just before TENS), at the 3rd hour (1 hour after the onset of TENS), at the 10th hour (just before the TENS), at the 11th hour (1 hour after the start of TENS), at the 18th hour ( Just before TENS) at the 19th Hour (1 hour after the start of TENS). TENS application hours will be arranged according to the patient in order to protect sleep integrity.
  Interventions: Other: Experimental group (Transcutaneous Electrical Nerve Stimulation)
- Control Group ( TENS will not be applied ) (No Intervention): Application of the control group: TENS will not be applied to this group.

INTERVENTIONS:
Other: Experimental group (Transcutaneous Electrical Nerve Stimulation) — The application will be applied at 8 hour intervals in the first 24 hours after the surgery.
  Arms: Experimental group ( TENS will be applied )

SUMMARY:
The aim of this study is to evaluate the effect of TENS (Transcutaneous Electrical Nerve Stimulation) on patient outcomes after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the standard treatment for symptomatic gallstones, acute cholecystitis and gallstone pancreatitis.Many complications can be seen after laparoscopic cholecystectomy.

The most common complication after laparoscopic cholecystectomy is pain. Pain appears as incisional, visceral and shoulder pain after laparoscopic cholecystectomy.After laparoscopic surgery, increased intra-abdominal pressure, stretching of the peritoneum, inability to take air given carbon dioxide (CO2), shoulder pain due to tension of muscle fibers due to diaphragm irritation, and visceral pain due to the interference of trocars on the abdominal wall as a result of intra-abdominal intervention are seen. After laparoscopic cholecystectomy, the effect of general anesthesia and the proximity of the incision area to the diaphragm may also cause pulmonary complications. Pneumoperiteneum developed by the administration of CO2 gas after laparoscopic cholecystectomy; Diaphragmatic irritation, increased intra-abdominal pressure, stretching of the peritoneum, and consequently the tension in the muscle fibers in the diaphragm can cause pain.

Inability to control pain can lead to many undesirable conditions in the patient, such as reluctance to mobilize, increased oxygen consumption, and delayed wound healing. This situation is also associated with increased hospital stay and financial burdens.In order to provide effective pain control, the combined use of pharmacological and non-pharmacological methods is important.Non-pharmacological methods are easy to learn, safe, have no definite contraindications, and provide pain management with non-drug applications. In a meta-analysis, it was determined that Transcutaneous Electrical Nerve Stimulation (TENS) is an effective, safe non-pharmacological method for symptomatic relief of pain and discomfort and no serious side effects were observed.

Studies have shown that TENS application reduces postoperative pain level and analgesia consumption. In addition, TENS application after laparoscopic cholecystectomy was found to be associated with a decrease in postoperative pain severity and complaints of nausea and vomiting. It is seen that there are not enough resources in the literature regarding the application of TENS after laparoscopic cholecystectomy.

The aim of this study is to evaluate the effect of TENS on patient outcomes after laparoscopic cholecystectomy.

.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Without pacemaker and arrhythmia,
* No previous history of chronic pain, alcohol or drug addiction,
* Not using TENS/opioids before surgery,
* Epidural analgesia is not applied in the postoperative period, without cognitive impairment,
* No thoracic incision other than cholecystectomy,
* Having at least 1 drain
* No metastatic disease
* No need for mechanical ventilation
* As a result of the evaluation by the physician, there is no objection to the application of TENS,
* Who agree to participate in the study,
* No postoperative complications
* Patients with American Society of Anesthesiology (ASA) evaluation I, II, III will be included in the sample group.

Exclusion Criteria:

* refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NRS) | 24 hours
  The scale ranges from 0 to 10. It is numbered from 0 to 10 according to the severity of the pain. 0 means no pain and 10 means the most severe pain.

SECONDARY OUTCOMES:
American Pain Society Patient Outcome | 24 hours
  American Pain Society Patient Outcome (APS-POQ) Questionnaire-Revised to measure pain management and patient satisfaction developed. (APS-POQ) is a tool designed to evaluate patients' experiences and satisfaction with pain management. Developed by the American Pain Society, the questionnaire aims to assess patient-centered outcomes in acute pain management.
  The scoring system of the APS-POQ varies depending on the version used and the study's objectives. However, in general, the items in the questionnaire assess various aspects of pain's impact, and lower scores typically indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cansel Bozer, Principal Investigator — Cukurova University
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir / Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No